CLINICAL TRIAL: NCT01571440
Title: The Effect of Soluble Corn Fiber on Calcium Utilization and Retention and Gut Microflora in Adolescents
Brief Title: Soluble Corn Fiber and Calcium Utilization in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Tate and Lyle Ingredients Americas LLC (Unknown)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Camp Calcium 11-Tate and Lyle
Record Dates: First submitted 2011-01-12; First posted 2012-04-05 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Osteoporosis
Keywords: Bone; adolescents; fiber; healthy; boys; girls; camp; calcium
MeSH Terms: conditions — Osteoporosis; Muscle Cramp

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Soluble Corn Fiber (Placebo Comparator): Each teen will receive a package of fruit snacks containing 0 g soluble corn fiber two times daily.
  Interventions: Dietary Supplement: No soluble corn fiber
- 12 g Soluble Corn Fiber (Active Comparator): Each teen will receive a package of fruit snacks containing 6 g soluble corn fiber two times daily
  Interventions: Dietary Supplement: 12 g soluble corn fiber

INTERVENTIONS:
Dietary Supplement: No soluble corn fiber — Each teen will receive a package of fruit snacks containing 0 g soluble corn fiber two times per day
  Other Names: soluble corn fiber
  Arms: No Soluble Corn Fiber
Dietary Supplement: 12 g soluble corn fiber — Each teen will receive a package of fruit snacks containing 6 g soluble corn fiber two times per day.
  Other Names: soluble corn fiber
  Arms: 12 g Soluble Corn Fiber

SUMMARY:
The purpose of this study was to determine the effect of soluble corn fiber on calcium absorption and retention and gut microflora in adolescent boys and girls.

DETAILED DESCRIPTION:
In a previous study, soluble corn fiber (SCF) was found to greatly enhance calcium utilization and bone properties in a growing rat model. Because factors that enhance bone density and mineral content can potentially result in a skeleton that will resist fracture later in life, it is important to investigate this potential in adolescents. Therefore, the objective of this study was to determine the effect of SCF on calcium absorption and retention in adolescent boys and girls. A second objective of this study was to assess whether additional dietary fiber leads to changes in gut microflora which may influence calcium absorption. During this two-phase metabolic camp participants consumed packages of fruit snacks supplemented with either 0 or 6 grams of soluble corn fiber twice a day during the first phase of the study, and switch to the opposite treatment during the second phase, with a 2-week washout period in between. Subjects collected all excreta during both phases and calcium absorption, gut microbiota, height, weight, and bone density were evaluated throughout the 6-week period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy, white adolescents (Hispanic or non-Hispanic)
* Boys age 13-15
* Girls age 12-14

Exclusion Criteria:

* Abnormal kidney or liver function
* Malabsorptive disorders
* Anemia
* Smoking
* History of medications that affect calcium metabolism
* Body weight outside 5-95 percentile body mass index (BMI) for age
* Regular consumption of illegal drugs
* Contraceptive use
* Pregnancy

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Calcium absorption and retention | up to three weeks
Gut microbial profile | up to three weeks

SECONDARY OUTCOMES:
Bone mineral content and density | up to three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Berdine Martin, PhD, Study Director — Purdue University; Connie Weaver, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States